CLINICAL TRIAL: NCT04873648
Title: The Effect of Intermittent Fasting Diet and Calorie-Restricted Diet on Dopamine and Serotonin Levels and Weight Management in Women With Obesity and Co-morbid Binge Eating Disorder and Food Addiction
Brief Title: Effect of Fasting and Calorie-Restricted Diets on Dopamine and Serotonin Levels Among Obese Women With BED and FA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, zainab zueter, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9/8/2020
Record Dates: First submitted 2021-04-27; First posted 2021-05-05 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Eating Disorders; Intermittent Fasting; Obesity
Keywords: Eating Disorders; Intermitted Fasting; Obesity; Dopamine; Serotonin
MeSH Terms: conditions — Feeding and Eating Disorders; Intermittent Fasting; Obesity | interventions — Therapeutics; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- food addiction and binge eating follow caloric reduced -intermitted fasting diet (Experimental): Obese women diagnosed with binge eating disorder and food addiction follow caloric reduced -intermitted fasting diet
  Interventions: Behavioral: caloric reduced -intermitted fasting diet
- food addiction and binge eating follow caloric restriction diet (Active Comparator): Obese women diagnosed with binge eating disorder and food addiction follow caloric restriction diet
  Interventions: Behavioral: Daily calorie restriction
- binge eating disorder follow follow caloric reduced -intermitted fasting diet (Experimental): Obese women diagnosed with binge eating disorder follow caloric reduced -intermitted fasting diet
  Interventions: Behavioral: caloric reduced -intermitted fasting diet
- binge eating disorder follow caloric restriction diet (Active Comparator): Obese women diagnosed with binge eating disorder follow a caloric restriction diet
  Interventions: Behavioral: Daily calorie restriction
- obese women without food addiction and binge eating follow caloric restriction diet (Placebo Comparator): Obese women without eating disorder follow a caloric restriction diet
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: caloric reduced -intermitted fasting diet — obese women with food addiction and binge eating follow intermittent calorie restriction diet ( time-restricted eating - typically 16 -hour fasting and 8-hour eating)
  Other Names: Treatment
  Arms: binge eating disorder follow follow caloric reduced -intermitted fasting diet; food addiction and binge eating follow caloric reduced -intermitted fasting diet
Behavioral: Daily calorie restriction — obese women with food addiction and binge eating disorder follow a Daily calorie restriction diet
  Other Names: Active comparative treatment
  Arms: binge eating disorder follow caloric restriction diet; food addiction and binge eating follow caloric restriction diet
Behavioral: Control group — obese women without food addiction and binge eating disorder follow a Daily calorie restriction diet
  Arms: obese women without food addiction and binge eating follow caloric restriction diet

SUMMARY:
Obesity presents a substantial economic burden in Jordan. Binge eating disorder (BED) and food addiction (FA) are the most common eating disorders associated with obesity. BED and FA most therapeutic approach is cognitive-behavioral therapy. Dopamine (DA) and serotonin (5HT) the major neurotransmitter responsible for FA and BED. Daily calorie restriction (CR) and intermittent calorie restriction (ICR) are two forms of diet therapy that can help weight loss. Prolong fasting increases lipolysis and elevates ketones bodies' levels in the brain led to a significant increase in the DA and 5HT. No prior human research has examined the effect of ICR (model 8:16) on DA and 5HT levels and weight reduction on obese with BED and FA. Therefore, A Randomized, controlled trial of 6 weeks follow-up will be used. A sample of 100 obese women will be selected to be randomly assigned to daily CR or ICR, or control group without FA or BED for a period of 6 weeks. Participants will be undergoing nutrition assessment, Anthropometrics assessment, food Addiction assessment (YFAS), binge eating assessment (BEDS-7), and hormonal level (DA&5HT) at baseline and after 6 weeks. The investigators anticipated that CR and ICR (model8:16) will significantly induce DA&5HT level changes and that ICR (model8:16) will be significantly more effective than CR in reducing BED & FA.

DETAILED DESCRIPTION:
This study will be conduct at nutritional and counseling center. This center is located at the south area of the city: Irbid- Jordan. It is licensed by the ministry of the health as a private nutritional center. This study has approval by Research Ethics Committee at the University of Jordan and by the Institutional Review Board (IRB) of Jordan University.

The present study is composed of 2 phases. In phase one random sample of two hundred (500) obese women aged 20-40 years will be selected initially to estimate the occurrence of binge eating disorder and food addiction. Phase two will be conducted on a nested sample of 100 obese women who selected to compare the effectiveness of dietary restriction versus intermittent fasting diet on weight reduction, hormonal changes among binge eaters and food addict women. These two groups will be compared with a control group (20 obese women without FA or BED).

The exclusion criteria will be as follows: subjects who get pregnant during the period of study, subjects with certain diseases such as chronic renal failure, chronic liver diseases, renal calculus, depression, subjects who were taking antidepressant drugs and any woman follows special diet Participants' information will be treated confidentially. However, only the researcher (PhD student) will know participants' names and she is the only one who will give them identification (ID) number The personal questionnaire will contain questions related to age, gender, education, employment, family income/month, residency area, smoking status, family history of FA, BED, depression, medications, previous and current health problems. As well as, questions about certain eating habits will be asked

Phase One:

A convenient sample of two 500 obese women aged 20-40 years who meets the inclusion criteria and agree to participate in the present study will be recruited in the present study. All selected sample will be assessed for BED and FA using the food Addiction assessment tool (YFAS), binge eating assessment (QEWP-5) .Also physical activity level will be assessed by GPPAQ (General Practice Physical Activity Questionnaire). Each subject will signed a consent form will be given an information sheet explaining the general background of the study regarding the research objectives Phase Two

The Intervention Procedure:

A Randomized, controlled trial of 6 weeks follow up will be conducted at the nutritional counseling center, Irbid, Jordan. A nested sample of 100 obese women will be selected to compare the effectiveness of dietary restriction versus intermittent fasting diet on weight reduction and hormonal changes among binge eaters and food addict women. After the completion of baseline measurement of anthropometric and biochemical data, subjects will be randomly assigned to daily calorie restriction (CR) or intermittent calorie restriction (ICR),or control group without FA or BED for a period of 6 weeks. All Subjects will follow the standard regimen that includes restricted calories diet, detailed individualized balanced menu (either regular diet or time restricted diet) based on the subject's baseline body weight and height. Macronutrient distribution of the assigned diets will provide carbohydrate (55-60%), protein (15-20%), fat (<30%). Instructions and counseling will be provided to all subjects individually; and they will be monitored every two weeks by the researcher. Each participant will be evaluated and monitored separately, and all information obtained will be confidential. Daily calorie requirements will be calculated using the Harris benedict equation for each subject, taking into consideration the activity level. About 1100 kcal/day deficit from initial energy body needs will be applied for each woman, and the expected calories content of the weight-reducing diets, which will be between 1200-1500 kcal/ day.

Women: (REE= 447.593 + 3.098 x (Ht cm) + 9.247 x (Wt kg) - 4.330 x (Age)) To monitor and evaluated the adherence of participants to their diet, they will be provide daily food record sheet, these sheet will be reviewed and discussed with the researcher.

Overnight fasting blood samples will be withdrawn from all groups before and after 6 weeks of the dietary intervention trial. Each time, a licensed Phlebotomist will collect about 20 mL of blood from each woman in tubes containing EDTA as anticoagulant. Samples then will be centrifuged immediately for 20 minutes at 2500 g at 4°C and plasma will be collected in 1.5 mL micro tubes and stored at -80°C until they were analyzed. Blood sample preparation and centrifugation will be performed by a specialist at the nutritional counseling center, Irbid, Jordan. The blood samples then will be transported and stored at -20°C until analyses in a private laboratory. Plasma samples will be assayed for dopamine and serotonin levels using sensitive ELISA kits for the quantification of Dopamine and serotonin.

ELIGIBILITY:
Inclusion Criteria:

* Females,
* Aged between 20-40 yr,
* Premenopausal,
* BMI(>30 kg/m)

Exclusion Criteria:

* Male
* Females aged <20-40< yr,
* Menopausal,
* BMI(<30 kg/m)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The most affected group with obesity and may have food Addiction and/or binge eating disorders
Enrollment: 100 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Dopamine serum level | Through study completion, an average of 1 year
  The level of serum dopamine in ng/ml at both baseline and 6 weeks of follow up
Serotonin serum level | Through study completion, an average of 1 year
  The level of serum serotonin in ng/ml at both baseline and 6 weeks of follow up
food addiction disorder | Through study completion, an average of 1 year
  by the diagnostic tool for food addiction - Yale Food Addiction Scale (YFAS), The content will be translated and the content validity will be assessed at both baseline and 6 weeks of follow-up. YFAS contains a 25-item self-report measure that includes mixed response categories (dichotomous and Likert-type format). The YFAS includes two scoring options: 1) a "symptom count" ranging from 0 to 7 that reflects the number of addiction-like criteria endorsed and 2) a dichotomous "diagnosis" that indicates whether a threshold of three or more "symptoms" plus clinically significant impairment or distress has been met. Food addiction can be "diagnosed" when three symptoms and clinically significant impairment or distress are present.
binge eating disorder (BED) | Through study completion, an average of 1 year
  by the diagnostic tool, to assess BED, a previously translated and validated eating and weight patterns questionnaire (QEWP-5) will be used based on the new diagnostic and statistical manual of mental disorders-5 criteria. at both baseline and 6 weeks of follow up The screening was based on the diagnostic criteria of the DSM-5 In the original form of the QEWP-5 questionnaire, if the participant answered based on the following criteria, the participant is considered to be diagnosed with BED.
  * 8 and 9 if the participant answered (YES) (Binge eating)
  * 10, 2, 3, 4, 5, or 6 (At least one episode per a week in the last 3 months)
  * 11 (a through e) 3 or more items marked "YES" (At least 3 associated symptoms during binge-eating episodes)
  * 13 (4 0R 5) (Marked distress regarding binge eating)

CONTACTS AND LOCATIONS:
Overall Officials: Rima H Mashal, Assoc. Prof, Study Chair — The University of Jordan
Locations (1):
- Zainb zaiter clinic, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The center (Jordan University hospital) where the study conducted emphasis of maintaining privacy and confidentiality of the participants' data

REFERENCES:
- [Background] Adams RC, Sedgmond J, Maizey L, Chambers CD, Lawrence NS. Food Addiction: Implications for the Diagnosis and Treatment of Overeating. Nutrients. 2019 Sep 4;11(9):2086. doi: 10.3390/nu11092086. PMID 31487791
- [Background] Ajlouni K, Jaddou H, Batieha A. Obesity in Jordan. Int J Obes Relat Metab Disord. 1998 Jul;22(7):624-8. doi: 10.1038/sj.ijo.0800637. PMID 9705020
- [Background] Allen GF, Ullah Y, Hargreaves IP, Land JM, Heales SJ. Dopamine but not l-dopa stimulates neural glutathione metabolism. Potential implications for Parkinson's and other dopamine deficiency states. Neurochem Int. 2013 Apr;62(5):684-94. doi: 10.1016/j.neuint.2012.12.004. Epub 2012 Dec 19. PMID 23261515
- [Background] Avena NM, Bocarsly ME, Hoebel BG, Gold MS. Overlaps in the nosology of substance abuse and overeating: the translational implications of "food addiction". Curr Drug Abuse Rev. 2011 Sep;4(3):133-9. doi: 10.2174/1874473711104030133. PMID 21999687
- [Background] Bastani A, Rajabi S, Kianimarkani F. The Effects of Fasting During Ramadan on the Concentration of Serotonin, Dopamine, Brain-Derived Neurotrophic Factor and Nerve Growth Factor. Neurol Int. 2017 Jun 23;9(2):7043. doi: 10.4081/ni.2017.7043. eCollection 2017 Jun 23. PMID 28713531
- [Background] Bello NT, Hajnal A. Dopamine and binge eating behaviors. Pharmacol Biochem Behav. 2010 Nov;97(1):25-33. doi: 10.1016/j.pbb.2010.04.016. Epub 2010 Apr 24. PMID 20417658
- [Background] Brownley KA, Berkman ND, Sedway JA, Lohr KN, Bulik CM. Binge eating disorder treatment: a systematic review of randomized controlled trials. Int J Eat Disord. 2007 May;40(4):337-48. doi: 10.1002/eat.20370. PMID 17370289
- [Background] Camandola S, Mattson MP. Brain metabolism in health, aging, and neurodegeneration. EMBO J. 2017 Jun 1;36(11):1474-1492. doi: 10.15252/embj.201695810. Epub 2017 Apr 24. PMID 28438892
- [Background] Citrome L. A primer on binge eating disorder diagnosis and management. CNS Spectr. 2015 Dec;20 Suppl 1:44-50; quiz 51. doi: 10.1017/S1092852915000772. PMID 26683528
- [Background] da Luz FQ, Hay P, Gibson AA, Touyz SW, Swinbourne JM, Roekenes JA, Sainsbury A. Does severe dietary energy restriction increase binge eating in overweight or obese individuals? A systematic review. Obes Rev. 2015 Aug;16(8):652-65. doi: 10.1111/obr.12295. Epub 2015 Jun 11. PMID 26094791
- [Background] Davis C. A commentary on the associations among 'food addiction', binge eating disorder, and obesity: Overlapping conditions with idiosyncratic clinical features. Appetite. 2017 Aug 1;115:3-8. doi: 10.1016/j.appet.2016.11.001. Epub 2016 Nov 2. PMID 27816464